CLINICAL TRIAL: NCT01745198
Title: Effect of Cerefolin®/CerefolinNAC® on Biomarker Measurements in Patients With Mild Cognitive Impairment, Alzheimer's Disease and Related Disorders
Brief Title: Effect of Cerefolin®/CerefolinNAC® on Biomarker Measurements
Status: Completed | Type: Observational
Sponsor: Pamlab, Inc. (Industry)
Collaborators: The Shankle Clinic (Unknown); Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Other Study IDs: NAC-002c
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Alzheimer's Disease Related Disorders
Keywords: homocysteinemia; dementia; depression; vitamin B12; folate; mild cognitive impairment; alzheimer's; homocysteine
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Homocysteinemia; Dementia; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A single blood draw for approximately 6-10 mL of blood will be performed for the total plasma homocysteine measurement and genetic studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment Group: This group consists of patients diagnosed with homocysteinemia who have been treated with Cerefolin®/CerefolinNAC® in the past or are currently being treated with Cerefolin®/CerefolinNAC®.
- Non-Treatment Group: This group consists of patients not diagnosed with homocysteinemia who have no past or current treatment with Vitamin B12, Folate or Cerefolin®/CerefolinNAC®.

SUMMARY:
In a retrospective analysis of data from 1100 patients, disease-delaying effects of Cerefolin®/CerefolinNAC® were examined in terms of cognition. The purpose of the current study is to expand the retrospective study dataset by prospectively collecting additional biomarker and imaging data.

DETAILED DESCRIPTION:
CerefolinNAC® is an orally administered prescription medical food, and is formulated as a combination of L-methylfolate calcium (as Metafolin®), methylcobalamin, and N-acetylcysteine. In a retrospective analysis, disease-delaying effects of Cerefolin®/CerefolinNAC® (CFLN) are examined in terms of cognition (measured by MCI Screen (MCIS)), and functional capacity (measured by Functional Assessment Staging Test (FAST)). - the treatment effect of CFLN on cognitive and functional measures, and on biomarker measures in patients with Alzheimer's disease and related disorders (ADRD).

The current study will expand the NAC-002b study dataset by prospectively collecting additional biomarker and imaging data in a more comprehensively assessed, matched sample of patients. This will allow more precise evaluation of cognitive and functional outcome measures, and biomarker measures will be assessed in an attempt to identify specific populations or conditions in which CFLN is most effective.

The sample will consist of patients with homocysteinemia plus past/current CFLN treatment (Treatment Group) matched to those without homocysteinemia plus no past/current B12, folate or CFLN treatment (Non-Treatment Group). Also 65 additional subjects will be recruited for the non-Treatment group, which will be used to improve the rate of decline estimates for the cognitive and functional outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of normal aging (NL), cognitive impairment or dementia not otherwise specified (CI/D), or ADRD
* With at least one previous quantitative MRI (qMRI)
* With at least one previous homocysteine level
* Without homocysteinemia plus no past or current B12, folate or Cerefolin® treatment, OR with homocysteinemia plus past or current Cerefolin® treatment

Exclusion Criteria:

Subjects who do not meet the inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with homocysteinemia plus past/current CFLN treatment (Treatment Group) will be matched to those without homocysteinemia plus no past/current B12, folate or CFLN treatment (Non-Treatment Group).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in rate of cognitive decline as measured by the Memory Performance Index (MPI) | Baseline to end of study (estimated average of 48 months)
  Change in MPI over time will be calculated using multiple retrospective time points.

SECONDARY OUTCOMES:
Change in rate of cognitive decline as measured by the MCI Screen | Baseline to end of study (estimated average of 48 months)
  Change in MCI Screen over time will be calculated using multiple retrospective time points.
Change in rate of cognitive decline as measured by The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Drawings | Baseline to end of study (estimated average of 48 months)
  Change in CERAD drawings over time will be evaluated using multiple retrospective time points
Change in rate of cognitive decline as measured by Trails A & B | Baseline to end of study (estimated average of 48 months)
  Change in Trails A & B over time will be assessed using multiple retrospective time points
Rate of atrophy of hippocampal volume | Baseline to end of study (estimated average of 48 months)
  Decrease in hippocampal volume over time will be assessed using volumetric MRI
Rate of atrophy in cortical volume | Baseline to end of study (estimated average of 48 months)
  Decrease in cortical volume over time will be assessed using volumetric MRI
Rate of atrophy in ventricular volume | Baseline to end of study (estimated average of 48 months)
  Decrease in ventricular volume over time will be assessed using volumetric MRI
Change in rate of cognitive decline as measured by Functional Assessment Staging Test (FAST) | Baseline to end of study (estimated average of 48 months)
  Change in FAST over time will be calculated using multiple retrospective time points.

CONTACTS AND LOCATIONS:
Overall Officials: William R Shankle, MS, MD, FACP, Principal Investigator — Shankle Clinic
Locations (1):
- Hoag Memorial Hospital, Newport Beach, California, United States